CLINICAL TRIAL: NCT05898750
Title: Antidiabetic Potential of Hyphanea Thebaica Fruits and Moringa Olifera Leaves
Brief Title: Antidiabetic Potiential of Moringa and Dom Extract
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Deraya University (Other)
Responsible Party: Principal Investigator, Soad Ali, Clinical professor, Deraya University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: MorDom
Record Dates: First submitted 2023-05-22; First posted 2023-06-12 (Actual); Last update posted 2023-09-26 (Actual); Status verified 2023-09

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental)
  Interventions: Dietary Supplement: MorDom
- Control group (No Intervention)

INTERVENTIONS:
Dietary Supplement: MorDom — oral powder in tea bags contains 4gm twice daily (equal concentration of each drugs)
  Arms: experimental group

SUMMARY:
The Antidiabetic potential of Hyphaene thebaica fruits and Moringa oleifera leaves will be investigated in diabetic patients (type 2). The patients will be maintained on tea of both drugs for 6 weeks. The fasting blood glucose levels of patients will be checked on a daily basis. Other blood biomarkers will be also reported such as insulin concentration, Lipid profile, liver enzymes, c-peptide and glycated hemoglobin

ELIGIBILITY:
Inclusion Criteria:

* diabetic patients type 2

Exclusion Criteria:

* liver failure
* heart failure
* renal failure

Ages: 30 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2023-04-22 (Actual); Primary Completion 2023-06-22 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Blood glucose level | 3 months
  measured by fast blood test

SECONDARY OUTCOMES:
blood level of lipid profile | two weeks
  Blood samples were drawn to measure levels of LDL, HDL, triglycerides, total cholesterol
Liver enzymes | two weeks
  Blood samples were drawn to measure levels of ALT and AST
C-peptide level | two weeks
  Blood samples were drawn to measure fasting and postprandial levels of c-peptide
Insulin level | two weeks
  Blood samples were drawn to measure fasting and postprandial levels of insulin

CONTACTS AND LOCATIONS:
Locations (1):
- Soad A. Mohamad, Minya, Egypt